CLINICAL TRIAL: NCT05269511
Title: Efficacy of Chinese Herbal Medicine to Prevent and Treat COVID-19 Close Contacts: A Randomized Controlled Trial
Brief Title: Efficacy of Chinese Herbal Medicine to Prevent and Treat COVID-19 Close Contacts
Acronym: CHM COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHM COVID-19
Record Dates: First submitted 2022-03-03; First posted 2022-03-08 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Chinese Herbal Medicine
  Interventions: Drug: Chinese herbal medicine is in the form of granules (9 g/sachet), which is comprised of ten medicinal herbs.
- Control group (No Intervention): usual care

INTERVENTIONS:
Drug: Chinese herbal medicine is in the form of granules (9 g/sachet), which is comprised of ten medicinal herbs. — Oral administration, twice per day.
  Other Names: Chinese herbal medicine
  Arms: Treatment group

SUMMARY:
This is a randomized, blank-controlled study in adults with household contact exposure to individuals with SARS-CoV-2 infection. All subjects in the study will be household contacts with close exposure to the first household member known to be newly infected with SARS-CoV-2. Subjects in each cohort will be randomly assigned to the Chinese herbal medicine treatment group or blank control group in a 4:1 ratio, followed by 1 week of the treatment period and 2 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Household contact exposure to individuals with SARS-CoV-2 infection
2. Aged ≥18
3. General healthy or have a chronic, stable medical condition
4. Voluntarily signing a written informed consent form
5. Able to follow written and oral instructions in Chinese

Exclusion Criteria:

1. Moderate to severe symptomatic SARS-CoV-2 infection
2. An allergic history to Chinese herbal drugs or a known allergy to the ingredients of the study drug
3. Pregnancy, breastfeeding or plan to become pregnant within the study timeframe
4. Vulnerable adults (i.e., mentally or physically disabled to take care of himself/herself)
5. Any physical examination findings, and/or history of any illness, or concomitant medications that, in the opinion of the study investigator, might not be suitable to participate in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2163 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who have PCR confirmed SARS-CoV-2 infection | 3 weeks
Proportion of subjects with treatment-emergent adverse events (TEAEs) and severity of TEAEs | 3 weeks
Proportion of subjects who subsequently develop COVID-19 symptoms or signs | 3 weeks
Proportion of subjects who subsequently develop moderate to severe COVID-19 infection | 3 weeks

SECONDARY OUTCOMES:
Number of days of symptomatic PCR confirmed SARS-CoV-2 infection | 3 weeks
Number of days of PCR confirmed SARS-CoV-2 infection | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Lyu, Study Director — School of Chinese Medicine, Hong Kong Baptist University
Locations (1):
- School of Chinese Medicine, Hong Kong Baptist University, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
All the individual participant data that underlie the results reported in the published article will be shared after de-identification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal

REFERENCES:
- [Derived] Du P, Lam WC, Leung C, Li H, Lyu Z, Yuen CS, Cheung CH, Lam TF, Bian Z, Zhong L. Efficacy and safety of Chinese herbal medicine to prevent and treat COVID-19 household close contacts in Hong Kong: an open-label, randomized controlled trial. Front Immunol. 2024 May 10;15:1359331. doi: 10.3389/fimmu.2024.1359331. eCollection 2024. PMID 38799438